CLINICAL TRIAL: NCT05538676
Title: Fluoride-labeled Boronophenylalanine PET Imaging in Patients With Solid Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiaohua Zhu (Other)
Responsible Party: Sponsor-Investigator, Xiaohua Zhu, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: 2022S150
Record Dates: First submitted 2022-08-24; First posted 2022-09-14 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Solid Tumor, Adult
Keywords: solid tumor BPA-PET

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: BPA-PET imaging — PET imaging

SUMMARY:
Recently, new high-dose radiation therapy [e.g., boron neutron capture therapy (BNCT)] absorbed into the tumor tissue has been applied to treat patients with solid tumors. Here we examine and describe how to evaluate the biological activity of tumors using positron emission tomography (PET) with fluoride-labeled boronophenylalanine (F-BPA) as a tracer.

DETAILED DESCRIPTION:
Boron Neutron Capture Therapy（BNCT） is an advanced cell-scale binary targeted radiotherapy technology that combines the advantages of targeted therapy and heavy ion therapy. BNCT provides a neutron source from a reactor or a medical accelerator. At the same time, the patient needs to be pre-injected with a boron-containing drug containing a non-radioactive boron 10 isotope. The boron drug enters the body and accumulates specifically in cancer cells. The patient receives epithermal neutron beam irradiation with high linear energy transfer (Linear EnergyTransferLET), thereby achieving the effect of killing tumor cells. Purpose，BNCT has more advantages over conventional radiotherapy, and normal tissue is better preserved than conventional radiotherapy.

PET imaging is a useful and effective technique to give absolute quantitative and biological distribution data of BPA in a non-invasive manner, and can add important characteristic parameters such as T/N ratio, SUV and Kinetic parameters. Given the complexity of BNCT, PET and PET/CT is currently the new standard for designing patient recruitment: The Methodology of L-18F-BPA PET is an important tool to design clinical trials , estimate the size of tumor and indicate the concentration ratio of BPA in surrounding normal tissues. Following this principle, researchers can accurately identify which patients can benefit from BNCT treatment through the selective accumulation of BPA in individual tumors. PET scans can provide a three-dimensional map of the boron distribution, which can be used for macroscopic dose calculations in the BNCT conventional neutron transmission code. Because most of the dose absorbed by living cells (65%) comes from the 10B(n,a)7Li response, the distribution of boron determines the variability of the main absorbed dose in the treatment plan. As a result, therapeutic schedule will be improved because the boron distribution will greatly affect the isodose line. Routine calculations provide a wider range of isodose contours, whereas PET produces contours that more closely approximate the observed clinical results of BNCT.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinically diagnosed solid tumors, including but not limited to recurrent head and neck cancer, glioma, pancreatic cancer, osteosarcoma, etc.; The selected subjects need to sign the informed consent.

Exclusion Criteria:

* Pregnant women; renal failure (serum Cr>3mg/dl); Patients with claustrophobia;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with diagnosed solid tumor
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-12-26 (Actual); Primary Completion 2023-08-25 (Estimated); Study Completion 2025-08-25 (Estimated)

PRIMARY OUTCOMES:
TBR（Tumor-to-Backgroud Ratio） | 1 year
  We delineate the region of interest (ROI), obtain the maximum standard uptake value (SUVmax) of the ROI in the PET/CT images. The target-to-background ratio (TBR) of the lesion was calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- TongjiHospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided